CLINICAL TRIAL: NCT06848751
Title: Non-intubated Thoracoscopic Surgery for Lung Leision in Patients With Impaired Pulmonary Function
Brief Title: Tubeless Surgery With Impaired Pulmonary Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRIP-ZYP
Record Dates: First submitted 2025-02-22; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Lung Function Decreased; Surgery
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tubeless group (Experimental): Non-intubated thoracoscopic surgery for lung leisions in patients with impaired pulmonary function
  Interventions: Procedure: Non-intubated thoracoscopic surgery

INTERVENTIONS:
Procedure: Non-intubated thoracoscopic surgery — Non-intubated thoracoscopic lung surgery for patients with impaired pulmonary function

SUMMARY:
Some patients with impaired lung function require minimally invasive surgical treatment, including those with lung cancer, benign lung tumors, pneumothorax, or lung volume reduction surgery. Patients with borderline lung function often cannot be extubated immediately postoperatively under conventional treatment models. These patients typically need to be transferred to the surgical ICU for close monitoring. However, positive-pressure mechanical ventilation with an endotracheal tube carries risks of further airway injury and persistent air leakage from the lung surface, leading to a high incidence of postoperative respiratory failure.

Non-intubated minimally invasive surgery (tubeless), which preserves spontaneous breathing without endotracheal intubation, avoids the physical stimulation of intubation and the airway damage caused by mechanical ventilation. This approach may reduce the incidence of postoperative airway injury and respiratory failure, potentially expanding the indications for minimally invasive lung surgery, lowering postoperative complication and mortality rates.

The aim is to further clarify the surgical indications for non-intubated single-port minimally invasive surgery in patients with impaired lung function, the decision-making criteria for postoperative ICU transfer, and the safety and feasibility of this comprehensive management approach.

DETAILED DESCRIPTION:
Research Background Some patients with impaired lung function require minimally invasive surgical treatment, including those with lung cancer, benign lung tumors, pneumothorax, or lung volume reduction surgery. After a thorough preoperative cardiopulmonary function assessment and multidisciplinary team (MDT) discussions, patients with borderline lung function often cannot be extubated immediately postoperatively under conventional treatment models. These patients typically need to be transferred to the surgical ICU for close monitoring. However, positive-pressure mechanical ventilation with an endotracheal tube carries risks of further airway injury and persistent air leakage from the lung surface, leading to a high incidence of postoperative respiratory failure.

Non-intubated minimally invasive surgery (tubeless), which preserves spontaneous breathing without endotracheal intubation, avoids the physical stimulation of intubation and the airway damage caused by mechanical ventilation. Throughout the procedure, patients maintain spontaneous breathing, and most can avoid ICU transfer postoperatively. Some patients may even be able to get out of bed on the same day of surgery. This approach may reduce the incidence of postoperative airway injury and respiratory failure, potentially expanding the indications for minimally invasive lung surgery, lowering postoperative complication and mortality rates, shortening hospital stays, and reducing costs and healthcare expenditures. It represents a new quality productivity in minimally invasive surgery.

Research Objectives The aim is to further clarify the surgical indications for non-intubated single-port minimally invasive surgery in patients with impaired lung function, the decision-making criteria for postoperative ICU transfer, and the safety and feasibility of this comprehensive management approach.

Research Methods

Literature Review: First, we will conduct a review of relevant medical literature to understand existing research outcomes and methodologies. This will provide a foundation and reference for our study.

Study Design: Based on the literature review, we will design a clinical trial for validation and exploration. This study is a prospective observational study aimed at confirming safety and feasibility while conducting exploratory analyses.

Data Analysis: Data obtained from the study will undergo statistical analysis and visualization to better interpret the experimental results. Appropriate statistical methods and software tools will be used to ensure data reliability and interpretability.

Expected Outcomes Through this study, we expect to define the surgical indications (lung function evaluation criteria and lung function improvement protocols) for non-intubated single-port minimally invasive lung resection in patients with impaired lung function. We aim to identify high-risk factors for postoperative ICU transfer and poor prognosis in these patients, thereby proposing a new safe protocol for minimally invasive surgery in this population. We hope to demonstrate the safety and efficacy of this approach, contributing to advancements in the medical field.

Research Significance The significance of this study lies in providing a new medical intervention protocol, offering a safe and effective comprehensive solution (including preoperative assessment, preoperative preparation, anesthesia and surgical interventions, and postoperative management) for minimally invasive lung resection in patients with impaired lung function. It addresses the current high-risk status of these patients undergoing surgery, potentially improving outcomes and reducing complications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with impaired lung function (who may require postoperative intubation and transfer to the surgical ICU after preoperative and MDT discussions).
2. Patients requiring minimally invasive lung resection due to lung cancer, pulmonary nodules, benign lung tumors, pneumothorax, lung volume reduction surgery, etc.
3. Patients with normal mental status who can cooperate with perioperative examinations, exercises, and physical rehabilitation measures.
4. Patients who agree to participate in the clinical trial after communication.

Exclusion Criteria:

1. Patients with severe impairment of cardiopulmonary function or other organ systems, who are deemed unable to tolerate any form of anesthesia or minimally invasive surgery after preoperative and MDT discussions.
2. Patients with abnormal mental status or who are unable to adequately cooperate with perioperative examinations, exercises, and physical rehabilitation measures.
3. Patients who refuse to participate in the clinical trial or decline the use of non-intubated anesthesia with preserved spontaneous breathing.
4. Patients who refuse to undergo surgery.

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
complication rate | within 30 days after surgery
  complication rate after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yunpeng Zhao, Principal Investigator — The Second Hospital of Shandong University
Locations (1):
- The Second Hospital of Shandong University, Jinan, Shandong, China